CLINICAL TRIAL: NCT06457932
Title: Effectiveness of Heart Rate Variability Biofeedback Training Versus a Meditation Program in Reducing Stress and Anxiety Levels in University Undergraduate Students.
Brief Title: Effectiveness of Heart Rate Variability Biofeedback Training Versus a Meditation Program in Reducing Stress Levels in University Undergraduate Students.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Hermann Fricke Comellas, PhD Student, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77859612N
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Stress; Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biofeedback training (Experimental): An 8-week intervention based on daily 10-minute HRV biofeedback training at rest using the Pulse HRV smartphone application.
  Interventions: Behavioral: Heart rate variability biofeedback training
- Meditation (Active Comparator): An 8-week intervention based on daily 10-minute guided meditation sessions led by an instructor with over 20 years of experience in teaching meditation.
  Interventions: Behavioral: Guided meditation
- Control (No Intervention): Passive, waitlist control group.

INTERVENTIONS:
Behavioral: Heart rate variability biofeedback training — An 8-week intervention based on daily 10-minute HRV biofeedback training at rest using the Pulse HRV smartphone application.
  Arms: Biofeedback training
Behavioral: Guided meditation — An 8-week intervention based on daily 10-minute guided meditation sessions led by an instructor with over 20 years of experience in teaching meditation.
  Arms: Meditation

SUMMARY:
The objective of this trial is to evaluate the efficacy of a heart rate variability biofeedback training protocol, compared to a guided meditation program and a control group, in reducing stress and anxiety levels among university undergraduate students.

ELIGIBILITY:
Inclusion Criteria:

1. Second- and third-year students of the Physiotherapy Degree at various universities in the province of Seville.
2. Enrolled in all courses for the academic year.
3. Enrolled in the courses for the first or second time.

Exclusion Criteria:

1. Having a job in addition to academic responsibilities.
2. Having a dependent family member under their care.
3. Diagnosed with any mental health issues.
4. Diagnosed with severe metabolic, cardiovascular, or respiratory conditions, or cancer.
5. Simultaneously pursuing another degree or a dual degree program.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Stress | T0: Before the intervention; T1: At one month, before the exam period; T2: At two months, after the semester ends; T3: At three-month follow-up
  Measured using the Percieved Stress Scale (PSS).
Anxiety State | T0: Before the intervention; T1: At one month, before the exam period; T2: At two months, after the semester ends; T3: At three-month follow-up
  Measured using the State-Trait Anxiety Inventory (STAI).

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | T0: Before the intervention; T1: At one month, before the exam period; T2: At two months, after the semester ends; T3: At three-month follow-up
  Measured using the Polar H10 band and Elite HRV app.
Academic Performance | T0: Before the intervention; T1: At one month, before the exam period; T2: At two months, after the semester ends; T3: At three-month follow-up
  Semester grade averages compared between groups.
Adherence | Daily during the 8 week intervention
  Tracked using an online calendar.

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Fricke-Comellas, PhD Student, Principal Investigator — University of Seville

IPD SHARING:
Plan to Share IPD: Undecided